CLINICAL TRIAL: NCT03595631
Title: Effects of Neurodynamic Interventions to Multimodal Physical Therapy in Patients With Multiple Sclerosis
Brief Title: Neurodynamic Interventions for Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Director of Department, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI-URJC 572
Record Dates: First submitted 2018-07-02; First posted 2018-07-23 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
Keywords: neurodynamics; pain
MeSH Terms: conditions — Multiple Sclerosis; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy (Active Comparator): Patients will receive 5 session of multimodal physiotherapy treatment of 30min duration including low-load strength exercises, soft tissue mobilization and muscle-tendon stretching exercises twice per week.
  Interventions: Other: Physical Therapy
- Physical Therapy plus neurodynamic (Experimental): Patients will receive 5 session of multimodal physiotherapy treatment of 30min duration including low-load strength exercises, soft tissue mobilization and muscle-tendon stretching exercises twice per week. In addition, they will also receive bilateral nerve slider neurodynamic interventions targeting the median, ulnar and radial nerves.
  Interventions: Other: Physical Therapy plus Neurodynamic

INTERVENTIONS:
Other: Physical Therapy — Patients will receive 5 session of multimodal physiotherapy treatment of 30min duration including low-load strength exercises, soft tissue mobilization and muscle-tendon stretching exercises twice per week.
  Arms: Physical Therapy
Other: Physical Therapy plus Neurodynamic — Patients will receive 5 session of multimodal physiotherapy treatment of 30min duration including low-load strength exercises, soft tissue mobilization and muscle-tendon stretching exercises twice per week. In addition, they will also receive bilateral nerve slider neurodynamic interventions targeting the median, ulnar and radial nerves.
  Arms: Physical Therapy plus neurodynamic

SUMMARY:
A randomized, parallel-group, clinical trial will be conducted to compare the immediate effects of the inclusion of a neurodynamic intervention into a multimodal physiotherapy program on pressure pain sensitivity, pain and manual dexterity in patients with multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of multiple sclerosis according to the modified McDonald criteria;
* symptoms of paresthesia and lack of sensitivity in the upper extremity;
* Expanded Disability Status Scale (EDSS) between 0 and 6.5 points;
* absence of cognitive deficit.

Exclusion Criteria:

* any exacerbation of multiple sclerosis during the previous 3 months;
* previous hand surgery or steroid injections treatment in the upper extremity;
* multiple diagnoses on the upper extremity (e.g., cervical radiculopathy);
* cervical, shoulder, or upper extremity trauma;
* other comorbid musculoskeletal medical conditions;
* mini-mental state examination <25

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Changes in pressure pain sensitivity | Baseline and one week after the last treatment session
  Pressure pain threshold over the median, ulnar and radial nerves, second metacarpal and tibialis anterior

SECONDARY OUTCOMES:
Changes in upper extremity pain intensity before and after the intervention | Baseline and one week after the last treatment session
  A Numerical Pain Rate Scale (NPRS, 0-10) will be used to record the mean and the worst intensity of pain in te upper extremity
Changes in light touch detection threshold | Baseline and after treatmentBaseline and one week after the last treatment session
  Light touch detection threshold will be assessed with a standardized set of modified twenty von Frey hairs
Changes in manual dexterity | Baseline and one week after the last treatment session
  Bilateral manual dexterity was bilaterally assessed using the nine-hole peg test

CONTACTS AND LOCATIONS:
Locations (1):
- César Fernández-de-las-Peñas, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Dios Perez-Bruzon J, Fernandez-de-Las-Penas C, Cleland JA, Plaza-Manzano G, Ortega-Santiago R. Effects of neurodynamic interventions on pain sensitivity and function in patients with multiple sclerosis: a randomized clinical trial. Physiotherapy. 2022 Jun;115:36-45. doi: 10.1016/j.physio.2021.04.004. Epub 2021 Apr 22. PMID 35101724